CLINICAL TRIAL: NCT07061145
Title: A Potential Relationship Between Treatment With Tyrosine Kinase Inhibitors and Erectile Dysfunction in Male Patients With Chronic Myeloid Leukemia
Acronym: ED2024
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 613/2024/OSS/IRCCSRE
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Myelocytic Leukemia; Erectile Dysfunctions; CVD - Cardiovascular Disease; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Erectile Dysfunction; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tirosin Kinase Inhibitors — Tyrosine kinase inhibitor (TKI) administered as part of standard clinical care for CML. No experimental treatment is applied. Exposure to the drug will be analyzed in association with erectile dysfunction outcomes.

SUMMARY:
Chronic myeloid leukemia (CML) is a myeloproliferative neoplasm characterized by the presence of the Philadelphia chromosome, resulting in the constitutive activation of the BCR-ABL1 tyrosine kinase. The advent of tyrosine kinase inhibitors (TKIs) has revolutionized the management of CML, trasforming it from a fatal disease to a chronic condition with excellent long-term outcomes for the majority of patients. The introduction of tyrosine kinase inhibitor (TKI) based treatment for CML has revolutionized the management of this previously fatal disease, achieving sustained disease-control in more than 90% of patients.

However, as patients with CML are often required to undergo lifelong TKI therapy to maintain disease control, concerns regarding the long-term safety and tolerability of these agents have emerged.

The efficacy of second and third-generation TKIs exceeds the efficacy of imatinib, owing to their potent impact on wild-type BCR-ABL1 and various BCR-ABL1 mutants, along with additional drug targets. Furthermore, TKIs exhibit activity on non-kinase targets (es. oxidoreductase NQO2 for nilotinib and imatinib).

The prolonged treatment duration and expanded TKIs repertoire have led the emergence of various unexpected non-hematologic adverse events (AE), notably vascular adverse events (VAEs).

Recent evidence indicates a relatively high incidence of severe arterial changes in TKI-treated patients, with VAEs frequency correlating with TKI dosage and treatment duration. However, data elucidating the clinical features of vascular events are lacking.

Hormonal alterations have been reported in patients treated with imatinib. The tyrosine-kinase receptors cKIT and PDGF receptors, along with their respective ligands, are expressed in the testis, where they play a role in stimulating testosterone secretion by Leydig cells. Prolonged imatinib use has been associated with reduced testosterone production due to PDGFR and cKit blockade in the testis, potentially leading to gynaecomastia in men.

Cardiovascular disease (CVD) remains the leading cause of mortality in the United States, accounting for nearly 40% of all deaths. CVD and ED share a variety of common risk factors, including hypertension, diabetes, dyslipidemia, smoking, obesity, physical inactivity, and metabolic syndrome. Screening and diagnosing ED hold significant potential for secondary prevention of CVD. Despite the estabilished association between ED and CVD, the precise mechanisms driving ED's predictive value for CVD are yet to be fully identified. Early deection and treatment of CVD during the critical time frame in which risk factors can be modified will effectively reduce the occurrence of fatal CV events in male patients with ED.

This is a multicentre national, retrospective, prospective, non-interventional study that focuses on male CML patients starting first-line treatment with TKIs between 1 January 2015 and 31 January 2022.

All enrolled patients will be involved in both retrospective and prospective evaluations.

The retrospective component of the study allows the collection of data on the onset of ED, documented in medical records, that occurred before enrolment. It also includes information from physical examinations and laboratory tests, such as complete blood count, serum biochemistry (including renal and liver function tests, lipid profile and glycosylated haemoglobin), molecular biology for BCR-ABL transcript levels and electrocardiography (ECG), collected retrospectively every six months from enrolment until the documented onset of ED. The prospective evaluation assesses the occurrence of ED in the six months prior to enrolment and during the two-year follow-up period.

The primary objective of the study is to assess the incidence of erectile dysfunction (ED) among male patients with chronic myeloid leukaemia (CML) undergoing treatment with tyrosine kinase inhibitors (TKIs), imatinib, dasatinib, nilotinib, bosutinib or ponatinib, focusing in particular on those individuals who report the appearance of associated symptoms after treatment.

DETAILED DESCRIPTION:
This is a multicenter, national, non-interventional observational study with both retrospective and prospective components. The study aims to assess the incidence and characteristics of erectile dysfunction (ED) in male patients with chronic-phase chronic myeloid leukemia (CML) treated with tyrosine kinase inhibitors (TKIs) - imatinib, dasatinib, nilotinib, bosutinib, or ponatinib - as frontline therapy.

Eligible patients are adult males (aged 18-75) who initiated TKI treatment between January 1, 2015, and January 31, 2022. Data will be collected from medical records (retrospective phase) and through a 24-month follow-up (prospective phase). The retrospective data include ED onset, clinical assessments, BCR-ABL levels, ECG, and laboratory results. The prospective phase monitors ED development, cardiovascular events, and potential ED resolution in patients achieving treatment-free remission.

The primary objective is to estimate the cumulative incidence of ED from the start of TKI therapy. Secondary objectives include evaluating potential associations between TKI type and ED, the link between ED and cardiovascular toxicity, and the reversibility of ED in patients discontinuing therapy.

Approximately 350 patients are expected to be enrolled. No additional diagnostic procedures are planned beyond standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic phase Philadelphia chromosome-positive (Ph+) and/or BCR-ABL-positive CML.
* Patients starting frontline treatment with TKIs between 01st January 2015 and 31st January 2022.
* Age greater than or equal to 18 years and not exceeding 75 years at the time of starting therapy.
* Male sex.
* Exposure to Hydroxyurea or Anagrelide before the initiation of TKI therapy is allowed
* Ability to provide informed consent, as demonstrated by a clear understanding of the study's objectives and procedures and the ability to make an informed and voluntary decision to participate
* Signed written informed consent according to ICH/EU/GCP and national and local laws.

Exclusion Criteria:

* Patients with advanced phases (accelerated or blastic phase) Ph+ and/or BCR-ABL+ CML
* Patients who experienced ED before TKI initiation

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult male patients (aged 18-75) diagnosed with chronic-phase Philadelphia chromosome-positive (Ph+) chronic myeloid leukemia (CML), who initiated frontline treatment with tyrosine kinase inhibitors (TKIs) between January 1, 2015, and January 31, 2022.
  Patients must not have experienced erectile dysfunction (ED) before TKI initiation. Both retrospective and prospective clinical data will be collected to assess the occurrence and characteristics of ED and related cardiovascular events.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence function (CIF) of ED | at 24 months
  The cumulative incidence function (CIF) of ED will be calculated from the date of first TKIs administration to the date of clinical evaluation of ED or end of follow-up, censored at the last available data. Interruptions of TKIs for causes other than ED will be considered competing risks, and CIF will be estimated by the Gooley method with 95% confidence intervals.
  ED will be assessed using the International Index of Erectile Function (IIEF-5) questionnaire, which ranges from 5 (worst) to 25 (best). Higher scores indicate better erectile function; a score of 21 or less generally indicates erectile dysfunction.
  This information, including the full scale name, range, and score interpretation, will be included in the trial documentation.

SECONDARY OUTCOMES:
Frequency of erectile dysfunction by type of TKI used (imatinib, dasatinib, nilotinib, bosutinib, ponatinib) | At t0, 6 months, 12 months, 18 months, 24 months
  The proportion of patients who experience ED will be analyzed according to the specific TKI used during the study period.
Frequency of ED resolution in patients who previously reported erectile dysfunction during TKI treatment | At t0, 6 months, 12 months, 18 months, 24 months
  In patients who develop ED during TKI treatment, resolution of symptoms will be tracked during follow-up to assess potential reversibility.
Incidence of cardiovascular toxicity in patients with ED during TKI treatment | At t0, 6 months, 12 months, 18 months, 24 months
  Cardiovascular adverse events will be recorded and analyzed in patients who develop ED during TKI treatment, to explore a potential association between ED and cardiovascular toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Capodanno, MD, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, RE, Italy